CLINICAL TRIAL: NCT04458805
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral NX-13 in Healthy Adult Male and Female Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Oral NX-13 in Healthy Adults Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Landos Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NX-13-1a
Record Dates: First submitted 2020-06-16; First posted 2020-07-07 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — NX-13

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, ascending dose, multi-cohort study. The study will be conducted in 2 parts: a single ascending dose (SAD) part (Part A) followed by a multiple ascending dose (MAD) part (Part B). The decision to escalate between dose levels and proceed to Part B will be based upon review of blinded available safety data by a Safety Review Committee.
  Part A: 35 healthy volunteers will be enrolled in a total of 5 cohorts. Each cohort will enroll 7 participants with 5 participants randomized to receive NX-13 and 2 participants randomized to receive placebo.
  Part B: 21 healthy volunteers will be enrolled in a total of 3 cohorts. Each cohort will enroll 7 participants with 5 participants randomized to receive NX-13 and 2 participants randomized to receive placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NX-13 250mg (Experimental): Dose escalation in Part A will be conducted in 5 cohorts (Cohorts 1 to 5). Seven participants will be enrolled in each cohort and randomized to receive either NX-13 or placebo (ratio 5:2). NX-13 will be administered to Cohort 1 participants at the starting dose of 250 mg and increased in each new cohort. Five nominal dose levels in the range of 250 to 4000 mg have been selected for evaluation in Part A. The starting dose level in Part B will be determined by the SRC based on safety and tolerability data obtained in Part A. A dose level will only be evaluated in Part B if determined to be safe and tolerable in Part A. It is anticipated that 3 dose levels will be evaluated in Part B in a total of 3 cohorts (Cohorts 6 to 8). Seven participants will be enrolled in each cohort and will be randomized to receive a single oral dose of either NX-13 or placebo (ratio 5:2), once daily for seven days. NX-13 dose levels to be evaluated in Part B will be in the range of 500 to 4000 mg.
  Interventions: Drug: NX-13 250 mg
- Placebo (Placebo Comparator): Dose escalation in Part A will be conducted in 5 cohorts (Cohorts 1 to 5). Seven participants will be enrolled in each cohort and randomized to receive either NX-13 or placebo (ratio 5:2). NX-13 will be administered to Cohort 1 participants at the starting dose of 250 mg and increased in each new cohort. Five nominal dose levels in the range of 250 to 4000 mg have been selected for evaluation in Part A. The starting dose level in Part B will be determined by the SRC based on safety and tolerability data obtained in Part A. A dose level will only be evaluated in Part B if determined to be safe and tolerable in Part A. It is anticipated that 3 dose levels will be evaluated in Part B in a total of 3 cohorts (Cohorts 6 to 8). Seven participants will be enrolled in each cohort and will be randomized to receive a single oral dose of either NX-13 or placebo (ratio 5:2), once daily for seven days. NX-13 dose levels to be evaluated in Part B will be in the range of 500 to 4000 mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NX-13 250 mg — Dose escalation in Part A will be conducted in a total of 5 cohorts (Cohorts 1 to 5). Seven participants will be enrolled in each cohort and will be randomized to receive either NX-13 or placebo (ratio 5:2). NX-13 will be administered to Cohort 1 participants at the starting dose of 250 mg. The NX-13 dose will be increased in each new cohort. Five nominal dose levels in the range of 250 to 4000 mg have been selected for evaluation in Part A.
  It is anticipated that 3 dose levels will be evaluated in Part B in a total of 3 cohorts (Cohorts 6 to 8). Seven participants will be enrolled in each cohort and will be randomized to receive a single oral dose of either NX-13 or placebo (ratio 5:2), once daily for seven days.
  Arms: NX-13 250mg
Drug: Placebo — Dose escalation in Part A will be conducted in a total of 5 cohorts (Cohorts 1 to 5). Seven participants will be enrolled in each cohort and will be randomized to receive either NX-13 or placebo (ratio 5:2). NX-13 will be administered to Cohort 1 participants at the starting dose of 250 mg. The NX-13 dose will be increased in each new cohort. Five nominal dose levels in the range of 250 to 4000 mg have been selected for evaluation in Part A.
  It is anticipated that 3 dose levels will be evaluated in Part B in a total of 3 cohorts (Cohorts 6 to 8). Seven participants will be enrolled in each cohort and will be randomized to receive a single oral dose of either NX-13 or placebo (ratio 5:2), once daily for seven days.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, ascending dose, multi-cohort study. The study will be conducted in 2 parts: a single ascending dose (SAD) part (Part A) followed by a multiple ascending dose (MAD) part (Part B).

The decision to escalate between dose levels and proceed to Part B will be based upon review of blinded available safety data by a Safety Review Committee.

DETAILED DESCRIPTION:
Part A: 35 healthy volunteers will be enrolled in a total of 5 cohorts. Each cohort will enroll 7 participants with 5 participants randomized to receive NX-13 and 2 participants randomized to receive placebo.

Part B: 21 healthy volunteers will be enrolled in a total of 3 cohorts. Each cohort will enroll 7 participants with 5 participants randomized to receive NX-13 and 2 participants randomized to receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers will be included in Part A or Part B of the study if they satisfy all the following criteria:

  1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects;
  2. Adult males and females, 18 to 64 years of age (inclusive) at screening;
  3. Body mass index (BMI) ≥ 19.0 and ≤ 31.0 kg/m2, with a body weight ≥ 60.0 and ≤ 85.0 kg at screening;
  4. Be nonsmokers (including tobacco, e-cigarettes and marijuana) for at least 1 month prior to first study drug administration;
  5. Medically healthy without clinically significant abnormalities at screening and pre-dose on Day 1, including:

     1. Physical examination without any clinically relevant findings;
     2. Systolic blood pressure in the range of 90 to 160 mmHg and diastolic blood pressure in the range of 50 to 95 mmHg after 5 minutes in supine position;
     3. Heart rate (HR) in the range of 50 to 100 bpm after 5 minutes rest in supine position;
     4. Body temperature, between 35.0°C and 37.5°C;
     5. No clinically significant findings in serum chemistry, hematology, coagulation and urinalysis tests as judged by the investigator;
  6. Conventional 12-lead ECG recording in triplicate (the mean of triplicate measurements will be used to determine eligibility at screening and Day-1) consistent with normal cardiac conduction and function, including:

     1. Normal sinus rhythm with HR between 50 and 100 bpm, inclusive;
     2. QTcF between 350 to 450 msec for male subjects and 350 to 470 msec for female subjects, inclusive;
     3. QRS duration of < 120 msec;
     4. PR interval of ≤ 210 msec;
     5. Electrocardiogram morphology consistent with healthy cardiac ventricular conduction and normal rhythm, and with measurement of the QT interval;
     6. No family history of short or long QT syndrome;
     7. No history of risk factors for torsade de pointes or the diagnosis;
  7. Female participants must: a. Be of nonchildbearing potential ie, surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause), or b. If of childbearing potential, must have a negative pregnancy test at screening (blood test) and before the first study drug administration (Day -1 urine test). They must agree not to attempt to become pregnant, must not donate ova, and must use a highly effective contraceptive method (Appendix 4) from signing the consent form until at least 30 days after the last dose of study drug.
  8. Male participants, if not surgically sterilized, must be willing not to donate sperm and, if engaging in sexual intercourse with a female partner who could become pregnant, must be willing to use a condom in addition to having the female partner use a highly effective contraceptive method (Appendix 4) from signing the consent form until at least 90 days after the last dose of study drug;
  9. Have suitable venous access for blood sampling;
  10. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

* Healthy volunteers will be excluded from Part A or Part B of the study if there is evidence of any of the following at screening, Day -1 or pre-dose on Day 1:

  1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past 3 months determined by the PI to be clinically relevant;
  2. Current infection that requires antibiotic, antifungal, antiparasitic or antiviral medications;
  3. Any history of malignant disease in the last 10 years (excludes surgically resected skin squamous cell or basal cell carcinoma);
  4. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia;
  5. Use of or plans to use systemic immunosuppressive (eg, corticosteroids, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (eg, interferon) during the study or within 4 months prior to the first study drug administration;
  6. Liver function test results (ie, AST, ALT, and gamma glutamyl transferase [GGT]) and total bilirubin must not be elevated more than 1.2-fold above the ULN;
  7. Positive test results for active human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies;
  8. History of active, latent or inadequately treated tuberculosis (TB) infection;
  9. Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs;
  10. Estimated creatinine clearance (CrCl) < 40 mL/min using the Cockcroft-Gault formula or serum creatinine more than 1.5-fold above the ULN;
  11. History of substance abuse or alcohol abuse within 12 months prior to first study drug administration;
  12. Positive drug or alcohol test results;
  13. Use of any prescription or over-the-counter medication (including herbal products, diet aids, and hormone supplements) within 10 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, except occasional use of paracetamol;
  14. Demonstrated clinically significant (required intervention, eg, emergency room visit, epinephrine administration) allergic reactions (eg, food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the investigator, would interfere with the volunteer's ability to participate in the trial;
  15. Known hypersensitivity to any of the study drug ingredients;
  16. Use of any live vaccinations within 30 days prior to the first study drug administration except for the influenza vaccine;
  17. For women of childbearing potential, a positive serum pregnancy test at screening or a positive urine pregnancy test with confirmatory serum pregnancy test on Day -1;
  18. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of first study drug administration;
  19. Participation in another investigational clinical trial within 60 days prior to the first study drug administration;
  20. Any other condition or prior therapy that in the opinion of the PI would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements;
  21. Is an employee of an investigator or sponsor or an immediate relative of an investigator.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Specific assessments to evaluate the incidence, severity and relationship of adverse events (AEs) | Part A: 37 days Part B: 44 days
  Specific assessments to evaluate treatment safety and tolerability include the following: the incidence, severity, and relationship of AEs
Incidence of abnormal Physical examination findings | Part A: 37 days Part B: 44 days
  Specific assessments to evaluate treatment safety and tolerability include the following: physical examinations
Measurement of body weight (Part B only) | Part A: 37 days Part B: 44 days
  Specific assessments to evaluate treatment safety and tolerability include the following: measurement of body weight (Part B only)
Incidence of abnormal clinical laboratory test results | Part A: 37 days Part B: 44 days
  Specific assessments to evaluate treatment safety and tolerability include the following: change from baseline in clinical laboratory parameters (ie, hematology, serum chemistry, coagulation, and urinalysis parameters)
Incidence of abnormal ECG results | Part A: 37 days Part B: 44 days
  Specific assessments to evaluate treatment safety and tolerability include the following: 12-lead ECG
Incidence of abnormal vital signs | Part A: 37 days Part B: 44 days
  Specific assessments to evaluate treatment safety and tolerability include the following: vital signs

SECONDARY OUTCOMES:
Plasma concentration of NX-13 | Part A: 37 days Part B: 44 days
  Blood samples for pharmacokinetic (PK) analysis will be collected prior to dosing and at several timepoints up to 48 hours post-dose. Plasma concentrations of NX-13 will be determined at each timepoint and used to calculate PK parameters.
Urine concentration of NX-13 | Part A: 37 days Part B: 44 days
  Urine samples for analysis of NX-13 concentrations may also be collected prior to dosing and within 0-48 hours post-dose.
Fecal concentration of NX-13 | Part A: 37 days Part B: 44 days
  Fecal samples for analysis of NX-13 concentrations may also be collected prior to dosing and within 24-48 hours post-dose.
Measurement of NX-13 levels in stool | Part A: 37 days Part B: 44 days
  A small stool sample will be collected pre and post-dose for the measurement of calprotectin in the feces.
  Changes in fecal calprotectin levels following administration of NX-13 will be evaluated. Elevated fecal calprotectin indicates the migration of neutrophils to the intestinal mucosa, which occurs during intestinal inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lichtiger, MD, Study Director — Landos Biopharma Inc.
Locations (1):
- Nucleus Network, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No